CLINICAL TRIAL: NCT01959529
Title: A Trial Comparing Cardiovascular Safety of Insulin Degludec Versus Insulin Glargine in Subjects With Type 2 Diabetes at High Risk of Cardiovascular Events
Acronym: DEVOTE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EX1250-4080; 2013-002371-17 (EudraCT Number); U1111-1141-7614 (Other: WHO); JapicCTI-142464 (Registry Identifier: JAPIC)
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin degludec (IDeg) (Experimental): All subjects will continue their current antidiabetic therapy except for the basal insulin component (if any) that will be replaced by the investigational product.
  Interventions: Drug: insulin degludec
- Insulin glargine (IGlar) (Active Comparator): All subjects will continue their current antidiabetic therapy except for the basal insulin component (if any) that will be replaced by the investigational product.
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin degludec — Injected once daily subcutaneously (s.c., under the skin)
  Arms: Insulin degludec (IDeg)
Drug: insulin glargine — Injected once daily subcutaneously (s.c., under the skin)
  Arms: Insulin glargine (IGlar)

SUMMARY:
This trial is conducted globally. The aim of this trial is to compare cardiovascular safety of insulin degludec versus insulin glargine in subjects with type 2 diabetes at high risk of cardiovascular events.

ELIGIBILITY:
Inclusion Criteria: - Type 2 diabetes - Age above or equal to 50 years with predefined previous cardiovascular disease(s) or renal disease or age above or equal to 60 years with predefined cardiovascular risk factors - HbA1c (glycosylated haemoglobin) above or equal to 7.0% or HbA1c below 7.0% and current insulin treatment corresponding to above or equal to 20 U of basal insulin per day - One or more oral or injectable antidiabetic agent(s) Exclusion Criteria: - An acute coronary or cerebrovascular event in the previous 60 days - Planned coronary, carotid or peripheral artery revascularisation - Chronic heart failure NYHA (New York Heart Association) class IV - Current or past (within the last 5 years) malignant neoplasms (except basal cell and squamous cell skin carcinoma)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7637 (Actual)
Dates: Start 2013-10-29 (Actual); Primary Completion 2016-10-16 (Actual); Study Completion 2016-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (348):
- United States (212):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Montgomery, Alabama
  - Novo Nordisk Investigational Site, Gilbert, Arizona
  - Novo Nordisk Investigational Site, Glendale, Arizona
  - Novo Nordisk Investigational Site, Litchfield Park, Arizona
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Little Rock, Arkansas
  - Novo Nordisk Investigational Site, Searcy, Arkansas
  - Novo Nordisk Investigational Site, Chula Vista, California
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Downey, California
  - Novo Nordisk Investigational Site, Duarte, California
  - Novo Nordisk Investigational Site, Encino, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Greenbrae, California
  - Novo Nordisk Investigational Site, Huntington Beach, California
  - Novo Nordisk Investigational Site, Inglewood, California
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, La Mesa, California
  - Novo Nordisk Investigational Site, Lancaster, California
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Los Alamitos, California
  - Novo Nordisk Investigational Site, Mission Hills, California
  - Novo Nordisk Investigational Site, Montclair, California
  - Novo Nordisk Investigational Site, Monterey, California
  - Novo Nordisk Investigational Site, North Hollywood, California
  - Novo Nordisk Investigational Site, Palm Springs, California
  - Novo Nordisk Investigational Site, Poway, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, San Ramon, California
  - Novo Nordisk Investigational Site, Santa Ana, California
  - Novo Nordisk Investigational Site, Sherman Oaks, California
  - Novo Nordisk Investigational Site, Thousand Oaks, California
  - Novo Nordisk Investigational Site, Tustin, California
  - Novo Nordisk Investigational Site, Ventura, California
  - Novo Nordisk Investigational Site, Vista, California
  - Novo Nordisk Investigational Site, Westminster, California
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, Golden, Colorado
  - Novo Nordisk Investigational Site, Danbury, Connecticut
  - Novo Nordisk Investigational Site, Norwalk, Connecticut
  - Novo Nordisk Investigational Site, Waterbury, Connecticut
  - Novo Nordisk Investigational Site, Boca Raton, Florida
  - Novo Nordisk Investigational Site, Boynton Beach, Florida
  - Novo Nordisk Investigational Site, Bradenton, Florida
  - Novo Nordisk Investigational Site, Brandon, Florida
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Cooper City, Florida
  - Novo Nordisk Investigational Site, Fleming Island, Florida
  - Novo Nordisk Investigational Site, Fort Lauderdale, Florida
  - Novo Nordisk Investigational Site, Gainesville, Florida
  - Novo Nordisk Investigational Site, Green Cove Springs, Florida
  - Novo Nordisk Investigational Site, Hialeah, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Naples, Florida
  - Novo Nordisk Investigational Site, New Port Richey, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Panama City, Florida
  - Novo Nordisk Investigational Site, Ponte Vedra, Florida
  - Novo Nordisk Investigational Site, Port Charlotte, Florida
  - Novo Nordisk Investigational Site, Port Orange, Florida
  - Novo Nordisk Investigational Site, South Miami, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Decatur, Georgia
  - Novo Nordisk Investigational Site, Dunwoody, Georgia
  - Novo Nordisk Investigational Site, Lawrenceville, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Savannah, Georgia
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Idaho Falls, Idaho
  - Novo Nordisk Investigational Site, Addison, Illinois
  - Novo Nordisk Investigational Site, Champaign, Illinois
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Crystal Lake, Illinois
  - Novo Nordisk Investigational Site, Gurnee, Illinois
  - Novo Nordisk Investigational Site, Hines, Illinois
  - Novo Nordisk Investigational Site, Springfield, Illinois
  - Novo Nordisk Investigational Site, Brownsburg, Indiana
  - Novo Nordisk Investigational Site, Evansville, Indiana
  - Novo Nordisk Investigational Site, Franklin, Indiana
  - Novo Nordisk Investigational Site, Greenfield, Indiana
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Michigan City, Indiana
  - Novo Nordisk Investigational Site, Muncie, Indiana
  - Novo Nordisk Investigational Site, Council Bluffs, Iowa
  - Novo Nordisk Investigational Site, Wichita, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Madisonville, Kentucky
  - Novo Nordisk Investigational Site, Monroe, Louisiana
  - Novo Nordisk Investigational Site, New Orleans, Louisiana
  - Novo Nordisk Investigational Site, Shreveport, Louisiana
  - Novo Nordisk Investigational Site, Slidell, Louisiana
  - Novo Nordisk Investigational Site, Bangor, Maine
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Watertown, Massachusetts
  - Novo Nordisk Investigational Site, Worcester, Massachusetts
  - Novo Nordisk Investigational Site, Ann Arbor, Michigan
  - Novo Nordisk Investigational Site, Buckley, Michigan
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, Kalamazoo, Michigan
  - Novo Nordisk Investigational Site, Livonia, Michigan
  - Novo Nordisk Investigational Site, Troy, Michigan
  - Novo Nordisk Investigational Site, Olive Branch, Mississippi
  - Novo Nordisk Investigational Site, Hazelwood, Missouri
  - Novo Nordisk Investigational Site, Jefferson City, Missouri
  - Novo Nordisk Investigational Site, Kansas City, Missouri
  - Novo Nordisk Investigational Site, Billings, Montana
  - Novo Nordisk Investigational Site, Kalispell, Montana
  - Novo Nordisk Investigational Site, Elkhorn, Nebraska
  - Novo Nordisk Investigational Site, Fremont, Nebraska
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, East Brunswick, New Jersey
  - Novo Nordisk Investigational Site, Hoboken, New Jersey
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Lake Success, New York
  - Novo Nordisk Investigational Site, Mineola, New York
  - Novo Nordisk Investigational Site, New Windsor, New York
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, North Massapequa, New York
  - Novo Nordisk Investigational Site, Northport, New York
  - Novo Nordisk Investigational Site, Rochester, New York
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Westfield, New York
  - Novo Nordisk Investigational Site, Asheville, North Carolina
  - Novo Nordisk Investigational Site, Burlington, North Carolina
  - Novo Nordisk Investigational Site, Cary, North Carolina
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Lexington, North Carolina
  - Novo Nordisk Investigational Site, Morehead City, North Carolina
  - Novo Nordisk Investigational Site, New Bern, North Carolina
  - Novo Nordisk Investigational Site, Statesville, North Carolina
  - Novo Nordisk Investigational Site, Whiteville, North Carolina
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Winston-Salem, North Carolina
  - Novo Nordisk Investigational Site, Fargo, North Dakota
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Delaware, Ohio
  - Novo Nordisk Investigational Site, Franklin, Ohio
  - Novo Nordisk Investigational Site, Maumee, Ohio
  - Novo Nordisk Investigational Site, Mentor, Ohio
  - Novo Nordisk Investigational Site, Perrysburg, Ohio
  - Novo Nordisk Investigational Site, Norman, Oklahoma
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Altoona, Pennsylvania
  - Novo Nordisk Investigational Site, Beaver, Pennsylvania
  - Novo Nordisk Investigational Site, Danville, Pennsylvania
  - Novo Nordisk Investigational Site, Hermitage, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Smithfield, Pennsylvania
  - Novo Nordisk Investigational Site, Uniontown, Pennsylvania
  - Novo Nordisk Investigational Site, Upper Darby, Pennsylvania
  - Novo Nordisk Investigational Site, Wilkes-Barre, Pennsylvania
  - Novo Nordisk Investigational Site, Anderson, South Carolina
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Moncks Corner, South Carolina
  - Novo Nordisk Investigational Site, Murrells Inlet, South Carolina
  - Novo Nordisk Investigational Site, Myrtle Beach, South Carolina
  - Novo Nordisk Investigational Site, Orangeburg, South Carolina
  - Novo Nordisk Investigational Site, Spartanburg, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Knoxville, Tennessee
  - Novo Nordisk Investigational Site, Memphis, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Tullahoma, Tennessee
  - Novo Nordisk Investigational Site, Arlington, Texas
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Carrollton, Texas
  - Novo Nordisk Investigational Site, Corpus Christi, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Fort Worth, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Humble, Texas
  - Novo Nordisk Investigational Site, Hurst, Texas
  - Novo Nordisk Investigational Site, Irving, Texas
  - Novo Nordisk Investigational Site, Lewisville, Texas
  - Novo Nordisk Investigational Site, Longview, Texas
  - Novo Nordisk Investigational Site, Lubbock, Texas
  - Novo Nordisk Investigational Site, Midland, Texas
  - Novo Nordisk Investigational Site, Odessa, Texas
  - Novo Nordisk Investigational Site, Pearland, Texas
  - Novo Nordisk Investigational Site, Richardson, Texas
  - Novo Nordisk Investigational Site, Round Rock, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Splendora, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Waco, Texas
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, Bennington, Vermont
  - Novo Nordisk Investigational Site, South Burlington, Vermont
  - Novo Nordisk Investigational Site, Midlothian, Virginia
  - Novo Nordisk Investigational Site, Norfolk, Virginia
  - Novo Nordisk Investigational Site, Richmond, Virginia
  - Novo Nordisk Investigational Site, Winchester, Virginia
  - Novo Nordisk Investigational Site, Richland, Washington
  - Novo Nordisk Investigational Site, Spokane, Washington
  - Novo Nordisk Investigational Site, Kenosha, Wisconsin
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Algeria (4):
  - Novo Nordisk Investigational Site, Algiers
  - Novo Nordisk Investigational Site, Constantine
  - Novo Nordisk Investigational Site, Oran
  - Novo Nordisk Investigational Site, Sidi Bel Abbes
- Argentina (5):
  - Novo Nordisk Investigational Site, CABA
  - Novo Nordisk Investigational Site, Córdoba
  - Novo Nordisk Investigational Site, Mar del Plata
  - Novo Nordisk Investigational Site, Rosario
  - Novo Nordisk Investigational Site, Zárate
- Brazil (8):
  - Novo Nordisk Investigational Site, Fortaleza, Ceará
  - Novo Nordisk Investigational Site, Brasília, Federal District
  - Novo Nordisk Investigational Site, Aparecida de Goiânia, Goiás
  - Novo Nordisk Investigational Site, Belém, Pará
  - Novo Nordisk Investigational Site, Mogi das Cruzes, São Paulo
  - Novo Nordisk Investigational Site, São Paulo, São Paulo
  - Novo Nordisk Investigational Site, Fortaleza
  - Novo Nordisk Investigational Site, Porto Alegre
- Canada (6):
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Winnipeg, Manitoba
  - Novo Nordisk Investigational Site, Chatham, Ontario
  - Novo Nordisk Investigational Site, Ottawa, Ontario
  - Novo Nordisk Investigational Site, Sarnia, Ontario
  - Novo Nordisk Investigational Site, Laval, Quebec
- Croatia (4):
  - Novo Nordisk Investigational Site, Bjelovar
  - Novo Nordisk Investigational Site, Osijek
  - Novo Nordisk Investigational Site, Slavonski Brod
  - Novo Nordisk Investigational Site, Zagreb
- Greece (2):
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Thessaloniki
- India (19):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Hyderbad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Ahmedabad, Gujarat
  - Novo Nordisk Investigational Site, Gurgaon, Haryana
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Kozhikode, Kerala
  - Novo Nordisk Investigational Site, Indore, Madhya Pradesh
  - Novo Nordisk Investigational Site, Goa, Maharashtra
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, New Dehli, New Delhi
  - Novo Nordisk Investigational Site, Bhubaneswar, Odisha
  - Novo Nordisk Investigational Site, Mohali, Punjab
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Coimbatore, Tamil Nadu
  - Novo Nordisk Investigational Site, Lucknow, Uttar Pradesh
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, Ludhiana
  - Novo Nordisk Investigational Site, New Delhi
- Italy (12):
  - Novo Nordisk Investigational Site, Bari
  - Novo Nordisk Investigational Site, Bergamo
  - Novo Nordisk Investigational Site, Catanzaro
  - Novo Nordisk Investigational Site, Chieti
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Milano (MI)
  - Novo Nordisk Investigational Site, Olbia
  - Novo Nordisk Investigational Site, Padua
  - Novo Nordisk Investigational Site, Palermo
  - Novo Nordisk Investigational Site, Ravenna
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Sesto San Giovanni (MI)
- Japan (8):
  - Novo Nordisk Investigational Site, Chuo-ku, Tokyo
  - Novo Nordisk Investigational Site, Kanagawa
  - Novo Nordisk Investigational Site, Kumamoto
  - Novo Nordisk Investigational Site, Miyazaki
  - Novo Nordisk Investigational Site, Nagano
  - Novo Nordisk Investigational Site, Ota-ku, Tokyo
  - Novo Nordisk Investigational Site, Ōta-ku
  - Novo Nordisk Investigational Site, Shinjuku-ku, Tokyo
- Malaysia (7):
  - Novo Nordisk Investigational Site, Alor Star
  - Novo Nordisk Investigational Site, Kota Samarahan
  - Novo Nordisk Investigational Site, Kuala Lumpur
  - Novo Nordisk Investigational Site, Kuantan
  - Novo Nordisk Investigational Site, Malacca
  - Novo Nordisk Investigational Site, Serdang
  - Novo Nordisk Investigational Site, Seremban
- Mexico (6):
  - Novo Nordisk Investigational Site, Guadalajara, Jalisco
  - Novo Nordisk Investigational Site, Cuernavaca, Morelos
  - Novo Nordisk Investigational Site, Distrito Federal, México, D.F.
  - Novo Nordisk Investigational Site, Aguascalientes
  - Novo Nordisk Investigational Site, Chihuahua City
  - Novo Nordisk Investigational Site, San Luis Potosí City
- Poland (8):
  - Novo Nordisk Investigational Site, Bytom
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Krakow
  - Novo Nordisk Investigational Site, Oświęcim
  - Novo Nordisk Investigational Site, Poznan
  - Novo Nordisk Investigational Site, Szczecin
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Zamość
- Romania (4):
  - Novo Nordisk Investigational Site, Alba Iulia, Alba
  - Novo Nordisk Investigational Site, Baia Mare, Maramureş
  - Novo Nordisk Investigational Site, Târgu Mureş, Mureș County
  - Novo Nordisk Investigational Site, Ploieşti, Prahova
- Russia (15):
  - Novo Nordisk Investigational Site, Kemerovo
  - Novo Nordisk Investigational Site, Kirov
  - Novo Nordisk Investigational Site, Krasnodar
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Nizhny Novgorod
  - Novo Nordisk Investigational Site, Rostov-on-Don
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Saratov
  - Novo Nordisk Investigational Site, Syktyvkar
  - Novo Nordisk Investigational Site, Tver'
  - Novo Nordisk Investigational Site, Tyumen
  - Novo Nordisk Investigational Site, Ulyanovsk
  - Novo Nordisk Investigational Site, Volgograd
  - Novo Nordisk Investigational Site, Yaroslavl
  - Novo Nordisk Investigational Site, Yekaterinburg
- South Africa (8):
  - Novo Nordisk Investigational Site, Port Elizabeth, Eastern Cape
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Pretoria, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, eMkhomazi, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Middleburg, Mpumalanga
  - Novo Nordisk Investigational Site, Brits, North West
  - Novo Nordisk Investigational Site, Cape Town, Western Cape
- South Korea (3):
  - Novo Nordisk Investigational Site, Goyang
  - Novo Nordisk Investigational Site, Seoul
  - Novo Nordisk Investigational Site, Suwon-si, Gyeonggi-do
- Spain (5):
  - Novo Nordisk Investigational Site, Granada
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valencia
- Thailand (4):
  - Novo Nordisk Investigational Site, Bangkok
  - Novo Nordisk Investigational Site, Bangkoknoi, Bangkok
  - Novo Nordisk Investigational Site, Chiang Mai
  - Novo Nordisk Investigational Site, Nakhon Ratchasima
- United Kingdom (8):
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Dundee
  - Novo Nordisk Investigational Site, Edinburgh
  - Novo Nordisk Investigational Site, Guildford
  - Novo Nordisk Investigational Site, Norwich
  - Novo Nordisk Investigational Site, Nuneaton
  - Novo Nordisk Investigational Site, Stevenage
  - Novo Nordisk Investigational Site, Wolverhampton

REFERENCES:
- [Background] Pollock RF, Heller S, Pieber TR, Woo V, Gundgaard J, Hallen N, Luckevich M, Tutkunkardas D, Zinman B; DEVOTE Study Group. Short-term cost-utility of degludec versus glargine U100 for patients with type 2 diabetes at high risk of hypoglycaemia and cardiovascular events: A Canadian setting (DEVOTE 9). Diabetes Obes Metab. 2019 Jul;21(7):1706-1714. doi: 10.1111/dom.13730. Epub 2019 Apr 14. PMID 30924579
- [Background] Pollock RF, Valentine WJ, Marso SP, Andersen A, Gundgaard J, Hallen N, Tutkunkardas D, Magnuson EA, Buse JB; DEVOTE study group. Long-term Cost-effectiveness of Insulin Degludec Versus Insulin Glargine U100 in the UK: Evidence from the Basal-bolus Subgroup of the DEVOTE Trial (DEVOTE 16). Appl Health Econ Health Policy. 2019 Oct;17(5):615-627. doi: 10.1007/s40258-019-00494-3. PMID 31264138
- [Result] Marso SP, McGuire DK, Zinman B, Poulter NR, Emerson SS, Pieber TR, Pratley RE, Haahr PM, Lange M, Frandsen KB, Rabol R, Buse JB. Design of DEVOTE (Trial Comparing Cardiovascular Safety of Insulin Degludec vs Insulin Glargine in Patients With Type 2 Diabetes at High Risk of Cardiovascular Events) - DEVOTE 1. Am Heart J. 2016 Sep;179:175-83. doi: 10.1016/j.ahj.2016.06.004. Epub 2016 Jun 18. PMID 27595693
- [Result] Marso SP, McGuire DK, Zinman B, Poulter NR, Emerson SS, Pieber TR, Pratley RE, Haahr PM, Lange M, Brown-Frandsen K, Moses A, Skibsted S, Kvist K, Buse JB; DEVOTE Study Group. Efficacy and Safety of Degludec versus Glargine in Type 2 Diabetes. N Engl J Med. 2017 Aug 24;377(8):723-732. doi: 10.1056/NEJMoa1615692. Epub 2017 Jun 12. PMID 28605603
- [Result] Zinman B, Marso SP, Poulter NR, Emerson SS, Pieber TR, Pratley RE, Lange M, Brown-Frandsen K, Moses A, Ocampo Francisco AM, Barner Lekdorf J, Kvist K, Buse JB; DEVOTE Study Group. Day-to-day fasting glycaemic variability in DEVOTE: associations with severe hypoglycaemia and cardiovascular outcomes (DEVOTE 2). Diabetologia. 2018 Jan;61(1):48-57. doi: 10.1007/s00125-017-4423-z. Epub 2017 Sep 15. PMID 28913575
- [Result] Pieber TR, Marso SP, McGuire DK, Zinman B, Poulter NR, Emerson SS, Pratley RE, Woo V, Heller S, Lange M, Brown-Frandsen K, Moses A, Barner Lekdorf J, Lehmann L, Kvist K, Buse JB; DEVOTE Study Group. DEVOTE 3: temporal relationships between severe hypoglycaemia, cardiovascular outcomes and mortality. Diabetologia. 2018 Jan;61(1):58-65. doi: 10.1007/s00125-017-4422-0. Epub 2017 Sep 15. PMID 28913543
- [Result] Pollock RF, Valentine WJ, Marso SP, Gundgaard J, Hallen N, Hansen LL, Tutkunkardas D, Buse JB; DEVOTE Study Group. DEVOTE 5: Evaluating the Short-Term Cost-Utility of Insulin Degludec Versus Insulin Glargine U100 in Basal-Bolus Regimens for Type 2 Diabetes in the UK. Diabetes Ther. 2018 Jun;9(3):1217-1232. doi: 10.1007/s13300-018-0430-4. Epub 2018 Apr 30. PMID 29713962
- [Result] Theilgaard H, Mollerup I, Helmark IC, Endahl L, Hoskin S, Hvelplund A, Amby LK, Moses AC. Developing, Planning and Conducting an Interim Analysis: Lessons From the DEVOTE Cardiovascular Outcomes Trial (Trial Comparing Cardiovascular Safety of Insulin Degludec Versus Insulin Glargine in Patients With Type 2 Diabetes at High Risk of Cardiovascular Events). Ther Innov Regul Sci. 2019 Mar;53(2):279-286. doi: 10.1177/2168479018776943. Epub 2018 May 24. PMID 29793353
- [Result] Brown-Frandsen K, Emerson SS, McGuire DK, Pieber TR, Poulter NR, Pratley RE, Zinman B, Ranthe MF, Gron R, Lange M, Moses AC, Orsy P, Buse JB; DEVOTE Study Group. Lower rates of cardiovascular events and mortality associated with liraglutide use in patients treated with basal insulin: A DEVOTE subanalysis (DEVOTE 10). Diabetes Obes Metab. 2019 Jun;21(6):1437-1444. doi: 10.1111/dom.13677. Epub 2019 Apr 1. PMID 30793465
- [Result] Pratley RE, Emerson SS, Franek E, Gilbert MP, Marso SP, McGuire DK, Pieber TR, Zinman B, Hansen CT, Hansen MV, Mark T, Moses AC, Buse JB; DEVOTE Study Group. Cardiovascular safety and lower severe hypoglycaemia of insulin degludec versus insulin glargine U100 in patients with type 2 diabetes aged 65 years or older: Results from DEVOTE (DEVOTE 7). Diabetes Obes Metab. 2019 Jul;21(7):1625-1633. doi: 10.1111/dom.13699. Epub 2019 Apr 15. PMID 30850995
- [Derived] Bergenstal RM, Hachmann-Nielsen E, Kvist K, Peters AL, Tarp JM, Buse JB. Increased Derived Time in Range Is Associated with Reduced Risk of Major Adverse Cardiovascular Events, Severe Hypoglycemia, and Microvascular Events in Type 2 Diabetes: A Post Hoc Analysis of DEVOTE. Diabetes Technol Ther. 2023 Jun;25(6):378-383. doi: 10.1089/dia.2022.0447. Epub 2023 May 8. PMID 37017470
- [Derived] Klein KR, Franek E, Marso S, Pieber TR, Pratley RE, Gowda A, Kvist K, Buse JB. Hemoglobin glycation index, calculated from a single fasting glucose value, as a prediction tool for severe hypoglycemia and major adverse cardiovascular events in DEVOTE. BMJ Open Diabetes Res Care. 2021 Nov;9(2):e002339. doi: 10.1136/bmjdrc-2021-002339. PMID 34819298
- [Derived] Amod A, Buse JB, McGuire DK, Pieber TR, Pop-Busui R, Pratley RE, Zinman B, Hansen MB, Jia T, Mark T, Poulter NR; DEVOTE Study Group. Risk factors for kidney disorders in patients with type 2 diabetes at high cardiovascular risk: An exploratory analysis (DEVOTE 12). Diab Vasc Dis Res. 2020 Nov-Dec;17(6):1479164120970933. doi: 10.1177/1479164120970933. PMID 33280425
- [Derived] Heller S, Lingvay I, Marso SP, Philis-Tsimikas A, Pieber TR, Poulter NR, Pratley RE, Hachmann-Nielsen E, Kvist K, Lange M, Moses AC, Andresen MT, Buse JB; DEVOTE Study Group. Risk of severe hypoglycaemia and its impact in type 2 diabetes in DEVOTE. Diabetes Obes Metab. 2020 Dec;22(12):2241-2247. doi: 10.1111/dom.14049. Epub 2020 Jul 9. PMID 32250536
- [Derived] Pratley RE, Husain M, Lingvay I, Pieber TR, Mark T, Saevereid HA, Moller DV, Zinman B; DEVOTE Study Group. Heart failure with insulin degludec versus glargine U100 in patients with type 2 diabetes at high risk of cardiovascular disease: DEVOTE 14. Cardiovasc Diabetol. 2019 Nov 15;18(1):156. doi: 10.1186/s12933-019-0960-8. PMID 31729990
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 438 sites in 20 countries as follows: Algeria: 6; Argentina: 4; Brazil: 10; Canada: 6; Croatia: 5; Greece: 6; India: 26; Italy: 10; Japan: 8; Republic of Korea: 4; Malaysia: 8; Mexico: 7; Poland: 8; Romania: 4; Russian Federation: 20; South Africa: 15; Spain: 6; Thailand: 6; United Kingdom: 8; United States: 271.
Groups:
- Insulin Degludec: Subjects received insulin degludec (IDeg) 100 units/mL once daily (OD) subcutaneously (S.C.; under the skin) in the thigh, upper arm, or the abdominal wall between dinner and bedtime. Subjects continued their pre-trial medication except for the basal insulin, which was replaced by investigational medicinal product (IMP; IDeg). The pre-trial bolus insulin was allowed and could be replaced with insulin aspart (IAsp) at the discretion of the investigator. For subjects previously receiving premixed/biphasic insulin the basal component was calculated and switched to IDeg OD, and the bolus insulin component to bolus insulin. For subjects previously receiving premixed/biphasic insulin twice daily (BID), the total basal component was calculated, reduced by 20- 30% and switched to IDeg OD, and the bolus component was calculated and switched to IAsp. The trial was event driven for with a realised observation period up to 33 months.
- Insulin Glargine: Subjects received insulin glargine (IGlar) 100 units/mL OD subcutaneously (S.C.; under the skin) in the thigh, upper arm, or the abdominal wall between dinner and bedtime. Subjects continued their pretrial medication except for the basal insulin, which was replaced by investigational medicinal product (IMP; IGlar). The pre-trial bolus insulin was allowed and could be replaced with IAsp at the discretion of the investigator. For subjects previously receiving premixed/biphasic insulin the basal component was calculated and switched to IGlar OD, and the bolus insulin component to bolus insulin. For subjects previously receiving premixed/biphasic insulin BID, the total basal component was calculated, reduced by 20- 30% and switched to IGlar OD, and the bolus component was calculated and switched to IAsp. The trial was event driven with a realised observation period up to 33 months.
Period: Overall Study
Arm/Group | Insulin Degludec | Insulin Glargine
Started | 3818 | 3819
Exposed | 3809 | 3806
Completed | 3742 | 3747
Not Completed | 76 | 72
Not completed — Adverse event (not hypoglycaemia) | 0 | 1
Not completed — Lost to Follow-up | 4 | 1
Not completed — Other | 70 | 68
Not completed — Hypoglycaemia | 1 | 1
Not completed — Lack of glycaemic control | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline analysis was based on the full analysis set (FAS), which included all randomised subjects.
Groups:
- Insulin Degludec: Subjects received IDeg 100 units/mL OD S.C. (under the skin) in the thigh, upper arm, or the abdominal wall between dinner and bedtime. Subjects continued their pre-trial medication except for the basal insulin, which was replaced by investigational medicinal product (IMP; IDeg). The pre-trial bolus insulin was allowed and could be replaced with IAsp at the discretion of the investigator. For subjects previously receiving premixed/biphasic insulin the basal component was calculated and switched to IDeg OD, and the bolus insulin component to bolus insulin. For subjects previously receiving premixed/biphasic insulin BID, the total basal component was calculated, reduced by 20- 30% and switched to IDeg OD, and the bolus component was calculated and switched to IAsp. The trial was event driven for with a realised observation period up to 33 months.
- Insulin Glargine: Subjects received IGlar 100 units/mL OD subcutaneously (S.C.; under the skin) in the thigh, upper arm, or the abdominal wall between dinner and bedtime. Subjects continued their pretrial medication except for the basal insulin, which was replaced by investigational medicinal product (IMP; IGlar). The pre-trial bolus insulin was allowed and could be replaced with IAsp at the discretion of the investigator. For subjects previously receiving premixed/biphasic insulin the basal component was calculated and switched to IGlar OD, and the bolus insulin component to bolus insulin. For subjects previously receiving premixed/biphasic insulin BID, the total basal component was calculated, reduced by 20- 30% and switched to IGlar OD, and the bolus component was calculated and switched to IAsp. The trial was event driven with a realised observation period up to 33 months.
- Total: Total of all reporting groups
Arm/Group | Insulin Degludec | Insulin Glargine | Total
Number analyzed (Participants) | 3818 | 3819 | 7637
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (7.3) | 65.0 (7.5) | 65.0 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1422 | 1437 | 2859
  Male | 2396 | 2382 | 4778
HbA1c [Mean (Standard Deviation); unit: percentage of HbA1c] | 8.44 (1.63) | 8.41 (1.67) | 8.43 (1.65)

OUTCOME MEASURES:

1. Primary Outcome: Time From Randomisation to First Occurrence of a Major Adverse Cardiovascular Event (MACE): Cardiovascular Death, Non-fatal Myocardial Infarction, or Non-fatal Stroke
Description: Time from randomisation to first occurrence of an event adjudication committee (EAC)-confirmed 3-component major adverse cardiovascular event (MACE): cardiovascular death, non-fatal myocardial infarction, or nonfatal stroke. Events with EAC-confirmed onset date between randomisation and individual end of trial were included in the analyses. The number of subjects experiencing first EAC-confirmed MACEs, date between randomisation to the end of trial, both days included were presented. The trial was event driven and planned to last up to a maximum of 60.5 months. The actual trial duration (time from first subject first visit to last subject last visit) was 35.6 months. The maximum trial duration for a single subject was 33.1 months.
Time Frame: From randomisation to individual end of trial date (maximum patient year observation: 2.75 years)
Population: The analysis was based on the FAS, which included all randomised subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec | Insulin Glargine
Number analyzed (Participants) | 3818 | 3819
Participants
  First EAC-confirmed MACE | 325 | 356
  Myocardial infarction (non-fatal) | 143 | 163
  Stroke (non-fatal) | 68 | 74
  Cardiovascular death | 114 | 119
Statistical Analysis 1: Comparison: Insulin Degludec vs Insulin Glargine; The hazard ratio (HR) (IDeg vs IGlar) was based on Cox regression with investigational medicinal product as only factor for primary analysis; Test type: Non-Inferiority — Non-inferiority of IDeg to IGlar was considered confirmed if the upper limit of the two-sided 95% confidence interval for the HR was below 1.3 or equivalent if the p-value for the one-sided test of null hypothesis (H0): HR≥1.3 against the alternative hypothesis (Ha): HR<1.3 was less than 2.5%; p < 0.001, Regression, Cox — p value : Refers to one-sided test of HR >= 1.3 (against Ha: HR<1.3); Hazard Ratio (HR) = 0.908, 95% CI 2-sided [0.781 to 1.055]

2. Secondary Outcome: Number of EAC-confirmed Severe Hypoglycaemic Episodes
Description: Number of severe hypoglycaemic episodes from week 0 to the last assessment (up to 35.6 months). The episode of severe hypoglycaemia is an episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions. The trial was event driven and planned to last up to a maximum of 60.5 months. The actual trial duration (time from first subject first visit to last subject last visit) was 35.6 months. The maximum trial duration for a single subject was 33.1 months.
Time Frame: From randomisation to individual end of trial (maximum patient year observation: 2.75 years)
Population: The analysis was based on the FAS, which included all randomised subjects.
Measure: Number; unit: Number of severe episodes
Arm/Group | Insulin Degludec | Insulin Glargine
Number analyzed (Participants) | 3818 | 3819
Number of severe episodes | 280 | 472
Statistical Analysis 1: Comparison: Insulin Degludec vs Insulin Glargine; Superiority was considered confirmed if the upper limit of the two-sided 95% confidence interval for the rate ratio (RR) was below 1.0 or equivalent if the p-value for the one-sided test of H0: RR ≥1.0 against Ha: RR <1.0, was less than 2.5%; Test type: Superiority; p < 0.001, Negative binomial regression — p-value : Refers to one-sided test of RR >= 1.0 (against Ha: RR<1.0); The model included treatment (IDeg vs IGlar) as a fixed factor and was fitted using the FAS; Rate ratio = 0.601, 95% CI 2-sided [0.476 to 0.759]

3. Secondary Outcome: Occurrence of at Least One EAC Confirmed Severe Hypoglycaemic Episode Within a Subject (Yes/no)
Description: Occurrence of at least one EAC-confirmed severe hypoglycaemic episode within a subject from week 0 to the last assessment (up to 35.6 months). The episode of severe hypoglycaemia is an episode requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions.
Time Frame: From randomisation to individual end of trial date (maximum patient year observation: 2.75 years)
Population: The analysis was based on the FAS, which included all randomised subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec | Insulin Glargine
Number analyzed (Participants) | 3818 | 3819
Participants | 187 | 252
Statistical Analysis 1: Comparison: Insulin Degludec vs Insulin Glargine; Superiority of IDeg to IGlar was considered confirmed if the upper limit of the two-sided 95% confidence interval for the odds ratio (OR) was below 1.0 or equivalent if the p-value for the one-sided test of H0: OR ≥1.0 against Ha: OR<1.0, was less than 2.5%; Test type: Superiority; p < 0.001, Regression, Logistic — p-value: Refers to one-sided test of OR >= 1.0 (against Ha: OR<1.0); The model was logistic regression with log-link function.The model included treatment (IDeg vs IGlar) as a fixed factor and was fitted using the FAS; Odds Ratio (OR) = 0.729, 95% CI 2-sided [0.600 to 0.866]

4. Secondary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Mean change in HbA1c from week 0 to month 24.
Time Frame: Randomisation to 24 months
Population: The analysis was based on the FAS. The number of subjects analysed are the number of subjects with the available data after 24 months.
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Insulin Degludec | Insulin Glargine
Number analyzed (Participants) | 2431 | 2404
percentage of HbA1c | -0.86 (1.51) | -0.84 (1.57)

ADVERSE EVENTS:
Time Frame: The adverse events were considered from the randomisation visit (week 0) to the follow up visit (end of treatment plus at least 30 days). The trial was event driven and planned to last up to a maximum of 60.5 months. The maximum trial duration for a single subject was 33.1 months.
Description: Safety was summarised using the FAS, which included all randomised subjects.
Arm/Group | Insulin Degludec | Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 1473/3818 | 1517/3819
Other Adverse Events (participants affected / at risk) | 0/3818 | 0/3819
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec (N=3818) | Insulin Glargine (N=3819)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal hernia obstructive (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Abdominal mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 10 (10) | 10 (10)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal panniculectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Abdominal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 2 (2) | 1 (1)
Abdominal wall haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal wall infection (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 5 (5)
Abscess rupture (Infections and infestations) | 0 (0) | 1 (1)
Abscess soft tissue (Infections and infestations) | 0 (0) | 1 (1)
Accelerated hypertension (Vascular disorders) | 4 (4) | 7 (7)
Accident at work (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Acid peptic disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 11 (12) | 8 (8)
Acute endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 1 (1) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 70 (79) | 95 (110)
Acute left ventricular failure (Cardiac disorders) | 7 (7) | 6 (6)
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 98 (111) | 115 (123)
Acute prerenal failure (Renal and urinary disorders) | 2 (2) | 2 (2)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6 (9) | 6 (6)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 24 (26) | 31 (35)
Acute stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 5 (5)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adult T-cell lymphoma/leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Affective disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 (1) | 2 (2)
Alcoholic liver disease (Hepatobiliary disorders) | 1 (1) | 0 (0)
Alcoholic pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 11 (12) | 34 (40)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anaesthetic complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anaesthetic complication pulmonary (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 1 (1) | 0 (0)
Anastomotic ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 36 (37) | 48 (53)
Angina unstable (Cardiac disorders) | 87 (94) | 79 (93)
Angioedema (Skin and subcutaneous tissue disorders) | 3 (4) | 8 (9)
Angiopathy (Vascular disorders) | 0 (0) | 1 (1)
Angioplasty (Surgical and medical procedures) | 2 (2) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Anuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2)
Aortic aneurysm (Vascular disorders) | 3 (3) | 3 (3)
Aortic aneurysm repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 3 (3) | 3 (3)
Aortic stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic valve disease (Cardiac disorders) | 3 (3) | 0 (0)
Aortic valve replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 7 (8) | 5 (5)
Aphasia (Nervous system disorders) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 4 (4) | 6 (6)
Appendix disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1) | 5 (5)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 2 (2)
Arteriogram coronary (Investigations) | 2 (2) | 2 (2)
Arteriosclerosis (Vascular disorders) | 3 (3) | 2 (2)
Arteriosclerosis coronary artery (Cardiac disorders) | 4 (4) | 7 (7)
Arteriosclerotic gangrene (Infections and infestations) | 0 (0) | 1 (1)
Arteriospasm coronary (Cardiac disorders) | 1 (1) | 0 (0)
Arteriovenous fistula operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 8 (9)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (8)
Arthritis bacterial (Infections and infestations) | 4 (4) | 3 (3)
Arthropathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 3 (3) | 5 (5)
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 8 (8)
Asthma-chronic obstructive pulmonary disease overlap syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 47 (55) | 56 (75)
Atrial flutter (Cardiac disorders) | 11 (11) | 6 (6)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 3 (3)
Atrioventricular block (Cardiac disorders) | 0 (0) | 3 (3)
Atrioventricular block complete (Cardiac disorders) | 6 (6) | 3 (3)
Atrioventricular block first degree (Cardiac disorders) | 2 (2) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 2 (2) | 1 (1)
Atrioventricular dissociation (Cardiac disorders) | 0 (0) | 2 (2)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Azotaemia (Renal and urinary disorders) | 2 (2) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
B-cell lymphoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Back disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 12 (12)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bacterial pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 1 (1)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 9 (9) | 7 (7)
Beta haemolytic streptococcal infection (Infections and infestations) | 1 (1) | 2 (2)
Bile duct adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 2 (2)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 1 (1)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Biopsy lung (Investigations) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 3 (3) | 3 (3)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder neck obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder outlet obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Bladder transitional cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Blindness (Eye disorders) | 0 (0) | 2 (2)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 2 (2)
Blood magnesium decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium decreased (Investigations) | 2 (2) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Blood pressure inadequately controlled (Vascular disorders) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brachial plexus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 8 (9) | 9 (9)
Brain injury (Nervous system disorders) | 3 (3) | 0 (0)
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Brain stem haemorrhage (Nervous system disorders) | 0 (0) | 2 (2)
Brain stem infarction (Nervous system disorders) | 2 (2) | 4 (4)
Brain stem stroke (Nervous system disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Breast cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast enlargement (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 16 (17) | 21 (21)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis viral (Infections and infestations) | 2 (2) | 2 (2)
Bundle branch block left (Cardiac disorders) | 2 (2) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1)
Cardiac ablation (Surgical and medical procedures) | 1 (1) | 2 (2)
Cardiac arrest (Cardiac disorders) | 26 (26) | 20 (21)
Cardiac complication associated with device (General disorders) | 1 (1) | 0 (0)
Cardiac death (General disorders) | 1 (1) | 2 (2)
Cardiac discomfort (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 24 (26) | 30 (33)
Cardiac failure acute (Cardiac disorders) | 7 (7) | 8 (8)
Cardiac failure chronic (Cardiac disorders) | 8 (12) | 10 (11)
Cardiac failure congestive (Cardiac disorders) | 134 (177) | 143 (206)
Cardiac hypertrophy (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac monitoring (Investigations) | 0 (0) | 1 (1)
Cardiac pacemaker battery replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1) | 1 (1)
Cardiac pacemaker replacement (Surgical and medical procedures) | 0 (0) | 4 (4)
Cardiac valve fibroelastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cardiac valve replacement complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 12 (12) | 9 (9)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 1 (1)
Cardiomegaly (Cardiac disorders) | 2 (2) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 4 (4) | 7 (7)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 2 (2)
Cardiorenal syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1)
Carotid artery disease (Nervous system disorders) | 2 (2) | 2 (2)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 3 (3)
Carotid artery stenosis (Nervous system disorders) | 15 (15) | 14 (15)
Cataract (Eye disorders) | 9 (13) | 3 (4)
Cataract diabetic (Eye disorders) | 1 (1) | 0 (0)
Cataract operation (Surgical and medical procedures) | 1 (1) | 1 (1)
Catheter site haematoma (General disorders) | 0 (0) | 1 (1)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Catheterisation cardiac (Investigations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 52 (64) | 61 (72)
Cellulitis orbital (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 2 (2)
Cellulitis streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 3 (3)
Cerebral arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 3 (3) | 4 (4)
Cerebral infarction (Nervous system disorders) | 5 (5) | 4 (5)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 11 (11) | 22 (23)
Cervical cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Cervical myelopathy (Nervous system disorders) | 2 (2) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervix haemorrhage uterine (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 2 (2) | 5 (5)
Chest pain (General disorders) | 16 (16) | 21 (22)
Chest wall abscess (Infections and infestations) | 1 (1) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 8 (8) | 4 (4)
Cholecystitis acute (Hepatobiliary disorders) | 6 (6) | 4 (4)
Cholecystitis chronic (Hepatobiliary disorders) | 3 (3) | 5 (5)
Cholecystitis infective (Infections and infestations) | 1 (1) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 8 (8) | 8 (8)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Chordae tendinae rupture (Cardiac disorders) | 0 (0) | 1 (1)
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Chronic hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 16 (18) | 26 (30)
Chronic left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 42 (54) | 56 (70)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 8 (8) | 4 (4)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Coagulation time prolonged (Investigations) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Colectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 6 (6) | 6 (6)
Colitis ischaemic (Gastrointestinal disorders) | 3 (6) | 2 (2)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colonic abscess (Infections and infestations) | 0 (0) | 1 (1)
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colostomy closure (Surgical and medical procedures) | 1 (1) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 2 (2)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 3 (3) | 4 (4)
Congenital ureterocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 3 (3) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Coombs negative haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cor pulmonale (Cardiac disorders) | 1 (1) | 2 (2)
Cor pulmonale acute (Cardiac disorders) | 1 (1) | 0 (0)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary artery bypass (Surgical and medical procedures) | 1 (1) | 2 (2)
Coronary artery disease (Cardiac disorders) | 80 (85) | 89 (91)
Coronary artery dissection (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery embolism (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery insufficiency (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 12 (12) | 5 (6)
Coronary artery restenosis (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 12 (12) | 5 (5)
Coronary ostial stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Coronary vascular graft occlusion (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Cranial nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1) | 2 (2)
Cyst (General disorders) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 3 (3)
Cystitis noninfective (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Dactylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Death (General disorders) | 27 (27) | 21 (21)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 13 (13) | 10 (10)
Dehydration (Metabolism and nutrition disorders) | 23 (23) | 16 (16)
Delirium (Psychiatric disorders) | 2 (2) | 5 (5)
Dementia (Nervous system disorders) | 2 (2) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 2 (2)
Dengue fever (Infections and infestations) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 5 (5) | 4 (4)
Depression suicidal (Psychiatric disorders) | 1 (1) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis infected (Infections and infestations) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 2 (2)
Device failure (Product Issues) | 1 (1) | 0 (0)
Device fastener issue (Product Issues) | 1 (1) | 0 (0)
Device inappropriate shock delivery (Product Issues) | 0 (0) | 1 (1)
Device lead damage (Product Issues) | 0 (0) | 1 (1)
Device loosening (Product Issues) | 0 (0) | 1 (1)
Device malfunction (Product Issues) | 1 (1) | 2 (3)
Device related infection (Infections and infestations) | 3 (3) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
Diabetic complication (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 10 (10) | 11 (11)
Diabetic foot infection (Infections and infestations) | 4 (4) | 8 (8)
Diabetic gangrene (Infections and infestations) | 0 (0) | 2 (2)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 5 (5) | 14 (14)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Diabetic mononeuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 3 (3)
Diabetic neuropathic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Diabetic retinopathy (Eye disorders) | 4 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 11 (14) | 3 (3)
Diastolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Diffuse large B-cell lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dilatation intrahepatic duct acquired (Hepatobiliary disorders) | 0 (0) | 1 (1)
Disseminated cryptococcosis (Infections and infestations) | 1 (1) | 0 (0)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 11 (13) | 14 (14)
Diverticulum (Gastrointestinal disorders) | 5 (5) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 7 (7) | 4 (4)
Drug administration error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 2 (2)
Dry gangrene (Vascular disorders) | 2 (2) | 1 (1)
Duodenal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal switch (Surgical and medical procedures) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal vascular ectasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 1 (1) | 1 (1)
Dysentery (Infections and infestations) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 17 (19)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Eczema infected (Infections and infestations) | 0 (0) | 2 (2)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram ST segment abnormal (Investigations) | 0 (0) | 1 (1)
Electrocardiogram ST segment elevation (Investigations) | 1 (1) | 0 (0)
Electrocardiogram ST-T change (Investigations) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Embolic cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 4 (4) | 2 (2)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Embolism arterial (Vascular disorders) | 0 (0) | 2 (2)
Embolism venous (Vascular disorders) | 1 (1) | 1 (1)
Empyema (Infections and infestations) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 6 (6) | 4 (4)
End stage renal disease (Renal and urinary disorders) | 12 (12) | 9 (9)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Endometrial hyperplasia (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocele (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enthesopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Epidural lipomatosis (Nervous system disorders) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Erosive duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 2 (2) | 2 (2)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Essential hypertension (Vascular disorders) | 1 (1) | 0 (0)
Essential tremor (Nervous system disorders) | 0 (0) | 1 (1)
Evans syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Exostosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
External ear cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Extra dose administered (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Extradural abscess (Infections and infestations) | 0 (0) | 2 (2)
Extremity necrosis (Vascular disorders) | 1 (1) | 3 (3)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Facial paralysis (Nervous system disorders) | 1 (1) | 1 (1)
Factor V deficiency (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 54 (57) | 55 (59)
Fatigue (General disorders) | 1 (1) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Fluid overload (Metabolism and nutrition disorders) | 4 (5) | 2 (5)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Foreign body reaction (General disorders) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 1 (1)
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gallbladder cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 5 (5) | 13 (16)
Gas gangrene (Infections and infestations) | 1 (2) | 0 (0)
Gastrectomy (Surgical and medical procedures) | 4 (4) | 3 (3)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric bypass (Surgical and medical procedures) | 3 (3) | 4 (4)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 2 (2) | 3 (3)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastritis (Gastrointestinal disorders) | 8 (8) | 6 (7)
Gastritis erosive (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastroduodenitis haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 13 (13) | 12 (12)
Gastroenteritis Escherichia coli (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 7 (7)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal angiodysplasia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 10 (10) | 15 (16)
Gastrointestinal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 (7) | 9 (10)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 4 (4) | 3 (3)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 2 (2)
Glaucoma (Eye disorders) | 1 (1) | 1 (1)
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 1 (1)
Gout (Metabolism and nutrition disorders) | 4 (4) | 7 (7)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Graft infection (Infections and infestations) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 1 (1)
H1N1 influenza (Infections and infestations) | 0 (0) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 1 (2) | 4 (4)
Haematuria (Renal and urinary disorders) | 2 (2) | 3 (3)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 3 (3)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 7 (7) | 9 (9)
Haemorrhagic arteriovenous malformation (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 3 (3) | 4 (4)
Haemorrhagic transformation stroke (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 4 (4) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 6 (6)
Heart valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 3 (3) | 2 (2)
Hemiplegic migraine (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Hepatic cirrhosis (Hepatobiliary disorders) | 3 (3) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 2 (2) | 3 (3)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic lesion (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatitis chronic active (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 4 (4)
Hepatorenal failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatorenal syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 3 (3) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 2 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Hydrocephalus (Nervous system disorders) | 1 (2) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 3 (3)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 11 (12) | 16 (16)
Hyperglycaemic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 18 (21) | 22 (24)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 17 (19) | 23 (24)
Hypertensive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 8 (8) | 8 (8)
Hypertensive emergency (Vascular disorders) | 3 (3) | 3 (3)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 4 (4)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 64 (77) | 49 (66)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 1 (2)
Hypoglycaemic seizure (Nervous system disorders) | 3 (5) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 27 (29) | 29 (33)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 8 (8) | 7 (7)
Hypotension (Vascular disorders) | 14 (14) | 14 (15)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (3)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (8)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
IIIrd nerve paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ilium fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 4 (5) | 7 (9)
Impaired healing (General disorders) | 1 (1) | 2 (2)
Implantable defibrillator insertion (Surgical and medical procedures) | 2 (2) | 1 (1)
Implantable defibrillator replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site infection (Infections and infestations) | 1 (1) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infected bite (Infections and infestations) | 0 (0) | 1 (1)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0)
Infected seroma (Infections and infestations) | 0 (0) | 1 (1)
Infected skin ulcer (Infections and infestations) | 3 (3) | 2 (2)
Infectious colitis (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 5 (5) | 3 (3)
Infusion site infection (Infections and infestations) | 0 (0) | 1 (2)
Inguinal hernia (Gastrointestinal disorders) | 3 (3) | 4 (4)
Inguinal hernia repair (Surgical and medical procedures) | 2 (2) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Inner ear disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Intensive care unit acquired weakness (Nervous system disorders) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional self-injury (Psychiatric disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 2 (2) | 6 (6)
International normalised ratio increased (Investigations) | 0 (0) | 2 (2)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 9 (9) | 3 (3)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 4 (4) | 2 (2)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 2 (2)
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intra-ocular injection (Surgical and medical procedures) | 1 (1) | 0 (0)
Intracardiac thrombus (Cardiac disorders) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 2 (2)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 5 (5)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 3 (3) | 7 (7)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Ischaemic hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Ischaemic limb pain (Vascular disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 43 (44) | 45 (50)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jejunostomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Joint abscess (Infections and infestations) | 1 (1) | 0 (0)
Joint arthroplasty (Surgical and medical procedures) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 4 (5) | 7 (8)
Knee operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 2 (2) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 3 (3) | 4 (4)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Lacunar infarction (Nervous system disorders) | 5 (5) | 2 (2)
Lacunar stroke (Nervous system disorders) | 1 (1) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 4 (4) | 3 (3)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lead dislodgement (Product Issues) | 1 (2) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 3 (3)
Left ventricular failure (Cardiac disorders) | 6 (7) | 3 (3)
Left ventricular hypertrophy (Cardiac disorders) | 1 (1) | 0 (0)
Leg amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leriche syndrome (Vascular disorders) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 3 (4) | 2 (2)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 1 (1)
Local swelling (General disorders) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 4 (4) | 3 (3)
Long QT syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 4 (4) | 4 (4)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 3 (3)
Lower limb fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 3 (3)
Lumbar radiculopathy (Nervous system disorders) | 2 (2) | 2 (2)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 12 (13) | 7 (7)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Lung adenocarcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1)
Lymphocele (Vascular disorders) | 0 (0) | 1 (1)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Macular fibrosis (Eye disorders) | 1 (1) | 2 (2)
Major depression (Psychiatric disorders) | 2 (2) | 2 (2)
Malignant hypertension (Vascular disorders) | 3 (3) | 5 (5)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Medical device site haemorrhage (General disorders) | 0 (0) | 1 (1)
Medical observation (Investigations) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Mental status changes (Psychiatric disorders) | 7 (7) | 8 (8)
Mesenteric haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mesothelioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 7 (7) | 9 (10)
Metabolic surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Microangiopathy (Vascular disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 3 (3) | 0 (0)
Migraine-triggered seizure (Nervous system disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 2 (2) | 2 (2)
Mononeuropathy multiplex (Nervous system disorders) | 0 (0) | 1 (1)
Motor neurone disease (Nervous system disorders) | 1 (1) | 0 (0)
Mucinous endometrial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mucormycosis (Infections and infestations) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 2 (2)
Multiple sclerosis relapse (Nervous system disorders) | 0 (0) | 1 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 48 (51) | 66 (68)
Myocardial ischaemia (Cardiac disorders) | 7 (7) | 9 (9)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Necrotising fasciitis (Infections and infestations) | 1 (1) | 0 (0)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 11 (11) | 9 (9)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrosclerosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 2 (2)
Nerve root compression (Nervous system disorders) | 1 (1) | 0 (0)
Neuroendocrine carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuropathic ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Neurotrophic keratopathy (Eye disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 47 (48) | 54 (63)
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-small cell lung cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 2 (2) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Obesity (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive shock (Vascular disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 3 (4)
Oedema due to cardiac disease (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 4 (4) | 4 (4)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 3 (3)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Oesophageal rupture (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 2 (2) | 2 (2)
Optic ischaemic neuropathy (Eye disorders) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 6 (6) | 8 (8)
Osteitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 32 (35) | 30 (31)
Osteogenesis imperfecta (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 20 (26) | 22 (23)
Osteomyelitis acute (Infections and infestations) | 1 (1) | 1 (1)
Osteomyelitis chronic (Infections and infestations) | 3 (3) | 4 (4)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 1 (2)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0)
Ovarian cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Pain (General disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 7 (8) | 5 (5)
Pancreatitis acute (Gastrointestinal disorders) | 6 (7) | 11 (16)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Paranoia (Psychiatric disorders) | 1 (1) | 0 (0)
Paraspinal abscess (Infections and infestations) | 1 (1) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1) | 4 (4)
Paronychia (Infections and infestations) | 1 (1) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Penile squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 2 (2) | 1 (2)
Peptic ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1) | 1 (1)
Perineal abscess (Infections and infestations) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 13 (13) | 12 (12)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 4 (4) | 4 (5)
Peripheral artery stenosis (Vascular disorders) | 2 (3) | 4 (4)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 3 (3) | 7 (7)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 2 (2)
Peripheral vascular disorder (Vascular disorders) | 11 (12) | 14 (17)
Peripheral venous disease (Vascular disorders) | 0 (0) | 2 (2)
Perirectal abscess (Infections and infestations) | 0 (0) | 2 (2)
Peritoneal abscess (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 2 (2) | 0 (0)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Personality change due to a general medical condition (Psychiatric disorders) | 1 (1) | 0 (0)
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 2 (2)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1)
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pilonidal cyst (Infections and infestations) | 0 (0) | 1 (1)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumatosis intestinalis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 90 (99) | 90 (102)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 4 (4)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 2 (2)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia staphylococcal (Infections and infestations) | 1 (1) | 2 (2)
Pneumonia streptococcal (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polyp (General disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Post procedural haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Post procedural infection (Infections and infestations) | 8 (8) | 2 (2)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Post procedural sepsis (Infections and infestations) | 0 (0) | 1 (1)
Post stroke depression (Psychiatric disorders) | 0 (0) | 1 (1)
Post-injection delirium sedation syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Postoperative abscess (Infections and infestations) | 3 (3) | 0 (0)
Postoperative fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative ileus (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 11 (12) | 2 (2)
Presyncope (Nervous system disorders) | 3 (3) | 12 (12)
Prinzmetal angina (Cardiac disorders) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 5 (5)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Prostate cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate infection (Infections and infestations) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Prostatitis Escherichia coli (Infections and infestations) | 0 (0) | 1 (1)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pseudohyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pseudomonal bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Pterygium (Eye disorders) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 10 (10)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 9 (9)
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 2 (2) | 4 (4)
Pulmonary veno-occlusive disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (2) | 11 (11)
Pyelonephritis acute (Infections and infestations) | 4 (4) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1)
Pyuria (Infections and infestations) | 0 (0) | 1 (1)
Radicular pain (Nervous system disorders) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 2 (2)
Radius fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 1 (1) | 1 (1)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3)
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Renal abscess (Infections and infestations) | 0 (0) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Renal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 14 (14) | 17 (17)
Renal impairment (Renal and urinary disorders) | 3 (3) | 4 (4)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal transplant failure (Immune system disorders) | 1 (1) | 0 (0)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Reperfusion injury (Vascular disorders) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 22 (23) | 18 (19)
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 1 (1)
Retinal vein occlusion (Eye disorders) | 1 (1) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 1 (1)
Retinopathy proliferative (Eye disorders) | 1 (1) | 0 (0)
Reversible ischaemic neurological deficit (Nervous system disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Rib fracture (Injury, poisoning and procedural complications) | 4 (4) | 2 (2)
Right ventricular failure (Cardiac disorders) | 2 (2) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 20 (21) | 18 (18)
Rotator cuff repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Roux loop conversion (Surgical and medical procedures) | 0 (0) | 1 (1)
Salivary gland calculus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Salivary gland mass (Gastrointestinal disorders) | 1 (1) | 0 (0)
Salpingitis (Infections and infestations) | 1 (1) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Schizoaffective disorder bipolar type (Psychiatric disorders) | 0 (0) | 1 (2)
Schizophrenia (Psychiatric disorders) | 3 (3) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 2 (2)
Seizure (Nervous system disorders) | 6 (8) | 6 (6)
Senile dementia (Nervous system disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 36 (37) | 31 (31)
Sepsis pasteurella (Infections and infestations) | 1 (1) | 0 (0)
Sepsis syndrome (Infections and infestations) | 1 (1) | 0 (0)
Septic arthritis staphylococcal (Infections and infestations) | 1 (1) | 1 (1)
Septic embolus (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 11 (11) | 12 (13)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 2 (2)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0)
Silent myocardial infarction (Cardiac disorders) | 4 (4) | 2 (2)
Sinus arrest (Cardiac disorders) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 3 (3)
Sinus node dysfunction (Cardiac disorders) | 6 (6) | 5 (5)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 2 (2)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 13 (13) | 6 (6)
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Small cell lung cancer extensive stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 9 (10) | 6 (6)
Social stay hospitalisation (Social circumstances) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 2 (2) | 0 (0)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Soft tissue sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Sphincter of Oddi dysfunction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Spigelian hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Spinal cord compression (Nervous system disorders) | 0 (0) | 2 (2)
Spinal decompression (Surgical and medical procedures) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fusion surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal laminectomy (Surgical and medical procedures) | 2 (2) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Spondylitic myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Stab wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stag horn calculus (Renal and urinary disorders) | 2 (2) | 0 (0)
Staphylococcal abscess (Infections and infestations) | 0 (0) | 2 (2)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 2 (2)
Staphylococcal infection (Infections and infestations) | 3 (3) | 5 (6)
Staphylococcal sepsis (Infections and infestations) | 2 (2) | 5 (5)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Steatohepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Stoma site reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 3 (3)
Streptococcal sepsis (Infections and infestations) | 3 (3) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 2 (2) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 2 (2) | 2 (2)
Subclavian steal syndrome (Vascular disorders) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 3 (3)
Subdiaphragmatic abscess (Infections and infestations) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 1 (1) | 3 (3)
Sudden death (General disorders) | 1 (1) | 8 (8)
Sudden hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 5 (6) | 3 (3)
Suicide attempt (Psychiatric disorders) | 0 (0) | 3 (3)
Superior vena cava stenosis (Vascular disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 4 (4) | 4 (4)
Surgical failure (General disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 25 (27) | 24 (29)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 2 (2) | 3 (3)
Systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 5 (5)
Temporal arteritis (Vascular disorders) | 1 (1) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Testicular seminoma (pure) stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thalamic infarction (Nervous system disorders) | 1 (1) | 3 (3)
Thalamus haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 4 (4) | 2 (4)
Thrombotic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 2 (2) | 0 (0)
Thyroidectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 1 (1) | 2 (2)
Toxic goitre (Endocrine disorders) | 0 (0) | 1 (1)
Toxic nodular goitre (Endocrine disorders) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 2 (2)
Transfusion-related acute lung injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transient global amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 28 (29) | 42 (44)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transurethral prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 1 (1)
Trifascicular block (Cardiac disorders) | 0 (0) | 2 (2)
Troponin increased (Investigations) | 1 (1) | 2 (2)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Tumour of ampulla of Vater (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Ulnar nerve palsy (Nervous system disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Umbilical hernia repair (Surgical and medical procedures) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 8 (8)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 5 (5)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ureteric injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 3 (3) | 5 (5)
Urethral stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 9 (9) | 2 (2)
Urinary tract infection (Infections and infestations) | 34 (37) | 30 (37)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 2 (3)
Urosepsis (Infections and infestations) | 10 (11) | 9 (9)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Uterine mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
VIth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vascular dementia (Nervous system disorders) | 1 (1) | 2 (2)
Vascular headache (Nervous system disorders) | 0 (0) | 1 (1)
Vascular insufficiency (Vascular disorders) | 0 (0) | 1 (3)
Vascular procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular stent restenosis (General disorders) | 3 (3) | 2 (3)
Vascular stent stenosis (General disorders) | 1 (1) | 0 (0)
Vascular stent thrombosis (General disorders) | 1 (1) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular fibrillation (Cardiac disorders) | 6 (7) | 5 (5)
Ventricular hypokinesia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 8 (9) | 12 (16)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 5 (5) | 3 (3)
Vertigo positional (Ear and labyrinth disorders) | 1 (1) | 3 (3)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Viraemia (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 3 (3)
Viral pericarditis (Infections and infestations) | 1 (1) | 0 (0)
Visual field defect (Nervous system disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (5) | 7 (7)
Vulval abscess (Infections and infestations) | 1 (1) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wound infection (Infections and infestations) | 2 (2) | 4 (4)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Wrong drug administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property"